CLINICAL TRIAL: NCT06152705
Title: Triple-blind Randomized Trial Comparing the Efficacy of fMRI-Guided vs. Standard iTBS in Treating Depression
Brief Title: Comparing the Efficacy of fMRI-Guided vs. Standard iTBS in Treating Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Sara Tremblay, Principal Investigator, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-019
Record Dates: First submitted 2023-09-18; First posted 2023-12-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depression; Depressive Disorder, Major; Depressive Episode
Keywords: fMRI; iTBS; neuronavigation
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study is a two-arm triple-blind randomized parallel assignment clinical trial as neither the participant, care provider, nor the outcomes assessor know the arm (or condition) assigned to the participants. There are two treatment "arms" in which half will receive fMRI navigated iTBS and the other half will receive neuronavigated iTBS determined by a study randomizer software.
  Master randomization list of treatment blinding will be kept by a scientist of the research centre that is not involved in the research project. This can be broken in case of emergency and they can then inform required medical professionals directly if necessary. Directly involved research staff will be blinded (including the PI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fMRI guided iTBS targetting (Experimental): The target selected is based on functional connectivity determined from the MRI scan.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Neuronavigation guided iTBS targetting (Active Comparator): A technique for treatment location targeting, based on structural images of the brain using standard coordinates.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a Health Canada approved treatment for major depression. Typical treatments involve 30 to 45 minutes daily sessions delivered over 4 to 6 weeks. Recent technical advances allowed the development of theta burst stimulation (TBS), a novel rTMS paradigm that reduces daily sessions to 3 to 4 minutes while maintaining the same clinical efficacy. This study will specifically be administering intermittent TBS (iTBS), which is a novel refinement of conventional rTMS and consists of bursts of 3 stimulations at 50 Hz at theta frequency (5 Hz).
  Other Names: rTMS; TMS; iTBS; TBS

SUMMARY:
In this triple-blind randomized controlled trial, we ask if targeting intermittent theta burst stimulation (iTBS) based on individual resting state connectivity improves treatment outcomes in major depressive disorder (MDD). For the trial, we will recruit 210 patients with major depressive disorder. Each patient will undergo a 30-40-minute MRI scan, after which they will receive a 6-week standard iTBS treatment. Participants will be randomized to receive iTBS either to the standard neuronavigated target (a technique for treatment location targeting, based on group-average connectivity) or to a personalized connectivity-guided target selected based on individual functional connectivity scans. The main outcome of this trial is response rate as determined by ≥ 50% reduction in Grid HRSD-17 scores. Secondary outcomes include remission rate, change in depression, anxiety and anhedonia symptoms, quality of life, and biological measures of heart rate variability, objective sleep measures and daily activity as a proxy of anhedonia - defined as a reduced ability to experience pleasure.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an FDA-approved and widely used focal, safe, well-tolerated, and non-invasive brain stimulation method for the treatment of depression, and has been approved in Canada. Typical clinical rTMS is delivered on the left dorsolateral prefrontal cortex (DLPFC) at a 10 Hz frequency over 30-45 minutes to induce an increase in cortical excitability, which outlasts the duration of stimulation. iTBS is a novel refinement of conventional rTMS. iTBS consists of bursts of 3 stimulations at 50 Hz at theta frequency (5 Hz). However, instead of 30 minute treatment sessions, iTBS has comparable clinical efficacy with only 3 minute treatment sessions. Currently roughly 50% of the people receiving rTMS treatment for depression respond to the treatment. One of the main goals of current research in rTMS is to find improvements in the protocol to increase the number of responders.

One of the potential ways to improve rTMS is to select the target based on individual resting state functional connectivity. Within the DLPFC, there are still several possible targets for the rTMS. Functional magnetic resonance imaging (fMRI) studies have shown that therapeutic effects of rTMS are related to its effects on the subgenual anterior cingulate cortex (sgACC; Broadman area 25). Past literature has shown that in MDD the effectiveness of a target is related to its connectivity with the sgACC. A recent study showed in a retrospective sample of MDD patients that response to rTMS correlates with the distance from the personalized connectivity-guided target rather than a group average target, opening the door for individualized connectivity-guided rTMS targeting. Yet, the question whether individualized connectivity-guided rTMS targeting improves rTMS outcomes in a prospective sample has never been investigated. In this two-arm triple-blind randomized parallel assignment clinical trial we will test if 6-week treatment using individualized connectivity-guided iTBS targeting leads to better outcomes in MDD compared to conventional neuronavigated iTBS.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study, participants must fulfill all the following criteria:

1. voluntary and competent to consent to study,
2. Adults aged 18 years old or older,
3. can speak and read English,
4. primary and/or predominant diagnosis of major depressive episode without psychotic features in the current episode (confirmed by a Mini-International Neuropsychiatric Interview),
5. depressive symptoms have not improved after ≥ 1 adequate dose of antidepressant trial in the current depressive episode,
6. moderate symptoms in the current depressive episode as indexed by a score of at least 15 on the Grid 17-item Hamilton Rating Scale for Depression (Grid HRSD-17),
7. have been referred to rTMS treatment by their treating physician, and took a free and informed decision to follow this treatment,
8. are able to adhere to treatment schedule,
9. have stable psychotropic medications (including prescribed cannabis) or psychotherapy regimen for at least four weeks prior to entering the trial,
10. have an education-adjusted score of ≥ 24 at the Mini-Mental State Evaluation (MMSE) if they are aged ≥ 65.

Exclusion criteria:

Participants fulfilling any of the following criteria will be excluded from the study:

1. diagnosis of bipolar I or II disorder, based on the DSM-5 criteria
2. current or past (< 3 months) substance (excluding caffeine or nicotine) or alcohol use disorder, as defined in DSM-5 criteria. Based on the DSM-5 criteria, mild cannabis or alcohol use disorder would be permissible in the past 3 months, moderate to severe would be an exclusion.
3. current use of illegal substances or cannabis (unless medical use, see note below), confirmed by urine drug screen
4. have a concomitant major unstable medical or neurologic illness (e.g. uncontrolled diabetes or renal dysfunction),
5. organic cause to the depressive symptoms (e.g. thyroid dysfunctions), as ruled out by the referring physician
6. acute suicidality or threat to life from self-neglect,
7. are pregnant or breastfeeding, or thinking of becoming pregnant during course of treatment (pregnancy will be assessed by a urine test),
8. have a specific contraindication for TMS (e.g., personal history of epilepsy or seizure, metallic head implant, pacemaker),
9. unwilling to maintain current antidepressant regimen,
10. are taking more than 1 mg of lorazepam per day or equivalent,
11. any other condition that, in the opinion of the investigators, would adversely affect the participant's ability to complete the study,
12. any contraindications for MRI
13. have failed a course of ECT within the current depressive episode due to the lower likelihood of response to rTMS (if they have had failed ECT in the past, this does not exclude them)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Compare the efficacy of fMRI guided TMS and conventional neuronavigated TMS on clinical response. | Administered at baseline (prior to first iTBS treatment) and every 2 weeks after that for 6 weeks (week 2, week 4, and week 6).
  Clinical response will be defined as a ≥ 50% reduction in the 17-Item Grid Hamilton Rating Scale for Depression (GRID-HRSD-17). The Grid HRSD is a clinician-rated instrument with seventeen items used to measure the severity of depressive episodes. Remission will be defined as a HRSD-17 score < 8 after 6 weeks of treatment.
  Score scale from 0 (better outcome, no depression thus better clinical response) to 60 (worst outcome, extreme depression thus worse clinical response).

SECONDARY OUTCOMES:
Change in severity of clinician-rated depressive symptoms as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS). | Administered at screening, before the first iTBS, week 2, week 4 and after iTBS treatment (week 6).
  As a secondary measure of depressive symptoms. Score scale from 0 (better outcome, no depression) to 52 (worst outcome, extreme depression).
Change in self-reported depression symptoms as measured by Beck Depression Inventory (BDI-II). | Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).]
  As a secondary measure of depressive symptoms. Score scale from 0 (better outcome, no depression) to 63 (worst outcome, extreme depression).
Change in self-reported anxiety symptoms as measured by Beck Anxiety Inventory (BAI) | Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).]
  As a secondary measure of anxiety symptoms. Score scale from 0 (better outcome, no depression) to 63 (worst outcome, extreme anxiety).
Change in self-reported suicidal thoughts symptoms as measured by Beck Scale for Suicidal Ideation (BSS). | Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).]
  To assess the effect of treatment on suicidal thoughts that may be improved by iTBS.
  Score scale from 0 (better outcome, no desire for suicide) to 38 (worst outcome, extreme desire for suicide).
Change in self-reported sleep quality as measured by Leeds Sleep Evaluation Questionnaire (LSEQ) | Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).]
  To assess the effect of treatment on self-report sleep that may be improved by iTBS.
  Score scale from 0 (better outcome, excellent sleep) to 100 (worst outcome, extremely poor sleep).
Change in self-reported sleep patterns as measured by Pittsburgh Sleep Quality Index (PSQI) | Before the first iTBS and after treatment (6 weeks).
  To assess the effect of treatment on self-report sleep that may be improved by iTBS.
  Score scale from 0 (better outcome, very high quality sleep) to 21 (worst outcome, very low quality sleep).
Change in quantity of sleep as measured with Empatica EmbracePlus Smartwatch | Start 2 weeks before the planned start date. Continuous measurement throughout study until the 2-week follow-up visit
  To assess the effect of treatment on objective measures of sleep patterns that may be improved by iTBS.
Change in perceived stress as measures with Perceived stress scale (PSS) | Administered at baseline before first iTBS treatment and after treatment completion (week 6).
  To assess the effect of treatment on self-report measures of stress that may be improved by iTBS.
  Score scale from 0 (better outcome, no perceived stress) to 40 (worst outcome, extreme perceived stress).
Change in physiological stress based on pulse rate and electrodermal activity response as measured with Empatica EmbracePlus Smartwatch | Start 2 weeks before the planned start date. Continuous measurement throughout study until the 2-week follow-up visit
  To assess the effect of treatment on objective measures of stress that may be improved by iTBS.
Change in self-reported anhedonia as measured by Snaith-Hamilton Pleasure Scale (SHAPS) | Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).]
  To assess the effect of treatment on self-report measures of anhedonia symptoms that may be improved by iTBS.
  Score scale from 0 (better outcome, no anhedonia) to 14 (worst outcome, extreme anhedonia).
Change in motion intensity (based on number of steps and total activity) as measured with Empatica EmbracePlus Smartwatch | Start 2 weeks before the planned start date. Continuous measurement throughout study until the 2-week follow-up visit.
  To assess the effect of treatment on objective measures of physical activity that may be improved by iTBS.
Change in motion heart rate variability as measured with Empatica EmbracePlus Smartwatch | Start 2 weeks before the planned start date. Continuous measurement throughout study until the 2-week follow-up visit.
  To assess the effect of treatment on objective measures of heart-rate variability, which has been shown to be linked to MDD and that may be improved by iTBS.
Change in self-reported hopelessness as measured by Beck Hopelessness Scale (BHS) | Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).
  To assess the effect of treatment on self-report symptoms of hopelessness that may be improved by iTBS.
  Score scale from 0 (better outcome, no sense of hopelessness) to 20 (worst outcome, extreme sense of hopelessness).
Change in quality of life as measured with Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Time Frame: Administered at baseline (prior to first iTBS treatment) and every week after that for 6 weeks (week 1, week 2, week 3, week 4, week 5, week 6).
  To assess the effect of treatment on self-report measures of quality of life that may be improved by iTBS.
  Score scale from 0 (worse outcome, poor life satisfaction and poor life quality) to 70 (better outcome, high life satisfaction and high quality of life).
Change in well-being as measured with Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS) | Administered before the first iTBS, week 2, week 4 and after iTBS treatment (week 6).
  To assess the effect of treatment on self-report measures of well-being that may be improved by iTBS.
  Score scale from 14 (worse outcome, poor mental wellbeing) to 70 (better outcome, excellent mental well).

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (6 weeks).
  Adverse events will be tracked and recorded.
Side Effects | Daily Monday-Friday throughout study (6 weeks).
  Side effects will be tracked and recorded on any TMS visits, using the TMS side effects questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tremblay, PhD, Principal Investigator — The Royal's Institute of Mental Health Research; Lauri Tuominen, MD PhD, Principal Investigator — The Royal's Institute of Mental Health Research
Locations (1):
- The Royal's Institute of Mental Health Research, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
After participants have completed their participation, we will ask them for informed consent for the storage of their de-identified data on OpenNeuro (an open access database) for the purpose of unspecified research for unspecified future research.
  If they do agree to participate, they will be given a unique study code (different from the participant ID used in the previous study) will be assigned to all of your study data instead of your personal identifying information (ex. 'John Smith' replaced by the unique study code 'A283422'). This unique study code will be used in the Open Access database to ensure your privacy and confidentiality (i.e. your de-identified study data cannot be linked to you in any way).
  In addition to an unique study code, their de-identified study data used in the Open Access database will include:
  * Age, sex, handedness, education level
  * Medical diagnosis and medication
  * Summary scores from clinical interviews
  * MRI scans
  * Treatment allocation
Supporting Information: SAP
Time Frame: Once your data has been included in the OpenNeuro database, your data cannot be removed or withdrawn as we will be unable to identify your information to separate it from the database.
Access Criteria: The shared data will hosted on the OpenNeuro (https://openneuro.org/) platform. The dataset becomes publically available under the Creative Commons Zero (CC0) Public Domain Dedication which places no restrictions on who can use the data or what can be done with them. The OpenNeuro is supported by the United States National Instututes of Mental Health BRAIN Initiative. The OpenNeuro follows the FAIR principles, which states that in order for shared data to be maximally useful for the scientific community, they need to be Findable, Accessible, Interoperable, and Reusable.
URL: https://openneuro.org/

REFERENCES:
- [Background] Mosimann UP, Schmitt W, Greenberg BD, Kosel M, Muri RM, Berkhoff M, Hess CW, Fisch HU, Schlaepfer TE. Repetitive transcranial magnetic stimulation: a putative add-on treatment for major depression in elderly patients. Psychiatry Res. 2004 Apr 30;126(2):123-33. doi: 10.1016/j.psychres.2003.10.006. PMID 15123391
- [Background] Shajahan PM, Glabus MF, Steele JD, Doris AB, Anderson K, Jenkins JA, Gooding PA, Ebmeier KP. Left dorso-lateral repetitive transcranial magnetic stimulation affects cortical excitability and functional connectivity, but does not impair cognition in major depression. Prog Neuropsychopharmacol Biol Psychiatry. 2002 Jun;26(5):945-54. doi: 10.1016/s0278-5846(02)00210-5. PMID 12369271
- [Background] Martin DM, McClintock SM, Forster J, Loo CK. Does Therapeutic Repetitive Transcranial Magnetic Stimulation Cause Cognitive Enhancing Effects in Patients with Neuropsychiatric Conditions? A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Neuropsychol Rev. 2016 Sep;26(3):295-309. doi: 10.1007/s11065-016-9325-1. Epub 2016 Sep 8. PMID 27632386
- [Background] Holtzheimer PE 3rd, Russo J, Claypoole KH, Roy-Byrne P, Avery DH. Shorter duration of depressive episode may predict response to repetitive transcranial magnetic stimulation. Depress Anxiety. 2004;19(1):24-30. doi: 10.1002/da.10147. PMID 14978782
- [Background] Avery DH, Holtzheimer PE 3rd, Fawaz W, Russo J, Neumaier J, Dunner DL, Haynor DR, Claypoole KH, Wajdik C, Roy-Byrne P. A controlled study of repetitive transcranial magnetic stimulation in medication-resistant major depression. Biol Psychiatry. 2006 Jan 15;59(2):187-94. doi: 10.1016/j.biopsych.2005.07.003. Epub 2005 Sep 1. PMID 16139808
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708